CLINICAL TRIAL: NCT04482608
Title: The Metastatic Colorectal Cancer Patients With Proficient Mismatch Repair (pMMR) / Microsatellite Stable (MSS) or Deficient Mismatch Repair (dMMR) / Microsatellite Instability High (MSI-H) Status Received Palliative Chemotherapy Efficacy and Survival
Brief Title: The mCRC Patients With pMMR/MSS or dMMR/MSI-H Status Received Palliative Chemotherapy Efficacy and Survival
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Clinical Professor, Sun Yat-sen University
Other Study IDs: dMMR/MSI-H and chemotherapy
Record Dates: First submitted 2020-07-18; First posted 2020-07-22 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer Metastatic; Mismatch Repair Deficiency; Microsatellite Instability High
Keywords: Colorectal Cancer Metastatic; Mismatch Repair Deficiency; Microsatellite Instability High; Chemotherapy
MeSH Terms: conditions — Turcot syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pMMR/MSS mCRC patients: The metastatic colorectal cancer patients with proficient mismatch repair or microsatellite stable status.
- dMMR/MSI-H mCRC patients: The metastatic colorectal cancer patients with deficient mismatch repair or microsatellite instability high status.

SUMMARY:
Deficient mismatch repair (dMMR) or microsatellite instability high (MSI-H) accounts for 4-5% in metastatic colorectal cancer (mCRC). The efficacy and survival of patients with dMMR/MSI-H status received palliative chemotherapy have not clear yet. In this study, the investigators observed the efficacy and survival of dMMR/MSI-H status mCRC patients received palliative first-line chemotherapy.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the one of most common cancer in the world. Loss of function of DNA mismatch repair (MMR) is an important mechanism of CRC development. Mutation or modification of MMR genes result in MMR protein deficient (dMMR) and microsatellite instability (MSI). It has been reported that the dMMR or MSI high (MSI-H) phenotype is present in approximately 15-18% of CRC patients. Most dMMR/MSI-H tumors are sporadic CRC, and only approximately 3% of dMMR/MSI-H tumors are Lynch syndrome (LS) or hereditary nonpolyposis colorectal carcinoma (HNPCC).

The dMMR/MSI-H status was reported to be a predictive marker for adjuvant chemotherapy. Multiple retrospective studies showed that dMMR/MSI-H is correlated with a favorable prognosis in stage II/III CRC. Previous studies suggested that dMMR/MSI status may be a predictive marker of decreased benefit form adjuvant monotherapy of 5-fluorouracil (5-FU) in patients with stage II disease, but not in those with stage III disease. For metastatic colorectal cancer (mCRC), the relationship of the MMR/MSI phenotype and prognosis is unclear. Some researchers found that CRC patients with the dMMR/MSI-H phenotype have a worse prognosis. But other researchers thought the dMMR/MSI-H phenotype is no associate to efficacy and survival of palliative chemotherapy, even is benefit for efficacy and survival.Therefore, the aim of this study was to clarify whether the status of dMMR/MSI-H affected progression-free survival (PFS) in mCRC patients who received first-line palliative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Histologically confirmed Metastatic colorectal adenocarcinoma;
3. Immunohistochemistry confirmed mismatch repair status or polymerase chain reaction (pCR) / next-generation sequencing (NGS) confirmed microsatellite status
4. Received palliative chemotherapy and have complete information of treatment

Exclusion Criteria:

1. Patients have not tested for mismatch repair or microsatellite
2. Patients have not received palliative chemotherapy or received palliative chemotherapy but treatment information incomplete

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The metastatic colorectal patients with different MMR or microsatellite status received palliative chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 671 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to 24-36 months
  PFS as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1

SECONDARY OUTCOMES:
Response rate | From first patient first visit to 6 month after last patient first visit
  Based on Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)
Disease Control Rate (DCR) | From first patient first visit to 6 month after last patient first visit
  Based on Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)
Overall survival | up to approximately 9 year
  The time from registration to death due to any cause, or censored at date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Jin, MD.,PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun yat-sen university cancer center, Guangzhou, Guangdong, China